CLINICAL TRIAL: NCT02400606
Title: The Effect of Constructing Versus Solving Virtual Patient Cases on Transfer of Learning: A Randomized Trial
Brief Title: The Effect of Constructing Virtual Patient Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Centre for Clinical Education (Unknown)
Responsible Party: Principal Investigator, Rikke Malene H. G. Jepsen, MD, PHD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H-1-2013-FSP-6
Record Dates: First submitted 2015-03-17; First posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: constructing VPs; knowledge and skills transfer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group were presented with a short case overview introducing four cardiopulmonary VP cases as well as the final diagnosis and had to complete the history, physical findings, and lab results, i.e. constructing VP cases.
  Interventions: Other: Constructing VP cases
- Control (Active Comparator): The participants were presented with a short case overview introducing four cardiopulmonary VP cases to be solved, i.e. solving VP cases.
  Interventions: Other: Solving VP cases

INTERVENTIONS:
Other: Constructing VP cases — The participants were presented with a short case overview. The control group solved the cases, whereas the intervention group also received the final diagnosis and had to complete the history, physical findings, and lab results. After a week, participants completed a transfer test involving two standardized patients presenting a respiratory case and a cardiology case, respectively. Performances were video-recorded and subsequently assessed by two blinded raters using the Reporter-Interpreter- Manager-Educator (RIME) framework. Knowledge gains were assessed using a pre- and post-test of a 95-item Multiple-Response-Questionnaire (MRQ).
  Arms: Intervention
Other: Solving VP cases — See above
  Arms: Control

SUMMARY:
The aim of the study was to explore the effect of actively constructing Virtual patient (VP) cases compared with solving VP cases using 'Web-SP', Stockholm University, Stockholm, Sweden on knowledge gains and skills transfer in a group of pre-clerkship medical students.

DETAILED DESCRIPTION:
Solving VP cases is associated with large improvements in learning but its effectiveness is dependent on active student involvement. Constructing VP cases rather than solving them may engage students more actively in encoding new information and integrating it with previous knowledge.

Fourth-year medical students were included and randomized to constructing (intervention) or solving (control) four cardiopulmonary VP cases. The participants were presented with a short case overview. The control group solved the cases, whereas the intervention group also received the final diagnosis and had to complete the history, physical findings, and lab results. After a week, participants completed a transfer test involving two standardized patients presenting a respiratory case and a cardiology case, respectively. Performances were video-recorded and subsequently assessed by two blinded raters using the Reporter-Interpreter- Manager-Educator (RIME) framework. Knowledge gains were assessed using a pre- and post-test of a 95-item Multiple-Response-Questionnaire (MRQ).

ELIGIBILITY:
Inclusion Criteria:

* fourth-year medical students, University of Copenhagen
* pre-study participation in the mandatory patient encounter skills course

Exclusion Criteria:

* medical students who had taken the three pre-clerkship years at other universities, because of curriculum discrepancies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the medical students' management of a simulated patient encounter using a RIME-structured scoring form | After working with the virtual patient cases for one week +/- 3 days
  The scoring form includes assessment on the roles Reporter, Interpreter, Manager and Educators and has been validated for patient encounters like described below. The requirements for the RIME elements have been defined in with a cardiology professor and a consultant respiratory physician.
  The medical students are exposed to two encounters with simulated patients after working with the virtual patients on their own. The students will obtain history and perform physical examination from the simulated patient for 15 minutes. The will be provided a journal form that can be quickly filled in, the patient encounter is video recorded. After this they have 20 minutes to write the journal in an electronic format.
  The video recorded patient encounter and the journal will be assessed by two physicians who have experience in rating medical students performance with the scoring form, the raters are blinded for if the students belong to the intervention arm of the study or not.

SECONDARY OUTCOMES:
Multiple Choice/Answers Questionnaire | When entering the study and after working with the virtual patient cases for one week +/- 3 days
  A delta value for the medical students' knowledge of respiratory medicine and cardiology after working with the virtual patients will be obtained. The students have been taught respiratory medicine, but not cardiology. Half the virtual patient cases the students have been working with are on respiratory medicine and the other half are on cardiology.
  The questionnaire has been checked by a cardiology professor and a consultant respiratory physician to ensure validity.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ringsted, MD MHPE PHD, Study Director — Centre for Clinical Education